CLINICAL TRIAL: NCT03305874
Title: Automated Prediction and Prevention of Contrast Induced Nephropathy After Cardiac Catheterization
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB17-1005
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Contrast-induced Nephropathy
Keywords: contrast-induced nephropathy (CIN); percutaneous coronary intervention (PCI); computer-based risk tool

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study Group: Prospectively, inpatients undergoing percutaneous coronary intervention (PCI) will be consented, and the computer-based contrast induced nephropathy (CBCIN) risk score will be calculated and displayed to the operator, along with suggested standard CIN-avoidance strategies during the PCI. Following the PCI, serum creatinine will be measured as per treating physician, but those who undergo at least two consecutive daily serum creatinine measurements starting the day after the procedure will be included in the study. These patients will be called 6 months and 12 months post-procedure to determine mortality and re-hospitalization status.
  Interventions: Other: Exposure to CBCIN risk score
- Comparator Group: Retrospectively, inpatients who underwent PCI and had at least two consecutive daily serum creatinine measurements will be selected. These patients will then be matched to the prospective patients, and matched by age and gender. Baseline CBCIN score will be calculated and other demographic and outcomes information will be obtained from medical records review.

INTERVENTIONS:
Other: Exposure to CBCIN risk score — The computer-based contrast induced nephropathy (CBCIN) risk score and associated standard hydration strategy will be displayed on a monitor in front of the treating interventional cardiologist during the entirety of the PCI case. Since this scoring system and hydration strategy are both available in the peer-reviewed literature, clinical use of these data and implementation of a CIN-avoidance strategy is not experimental; however, the display of these data to interventional cardiologists is experimental. Based on exposure to these data, the treating interventional cardiologist may use the information as clinically appropriate (i.e. it is not the basis for clinical decisions).
  Groups: Study Group

SUMMARY:
Contrast agent is typically used during routine cardiac intervention in order to enhance the imaging necessary to perform the procedure. Using this contrast agent could lead to kidney injury, called contrast induced nephropathy (CIN). Currently, the methods used to reduce the risk of CIN include reducing the amount of contrast agent used and using a hydration strategy during procedure. A computer-based risk tool has been developed which reports a risk score for the likelihood a person undergoing cardiac intervention gets CIN and a proposed corresponding hydration strategy to reduce the risk of CIN. The purpose of this study is to determine whether the rate of CIN decreases when the treating physician has access to this risk tool during the procedure.

DETAILED DESCRIPTION:
This is a case-control series comparing a strategy using a computer-based contrast induced nephropathy (CBCIN) risk tool in patients undergoing PCI versus usual care. Only inpatients will be included in this study. These inpatients will be compared to historical controls obtained using the medical record of age- and gender-matched inpatients who underwent cardiac catheterization with at least two consecutive daily post-procedure creatinine values. The percentage PCI will be matched in the retrospective series.

In the prospective group, the operator will be exposed to the CBCIN risk tool before and during care delivery with estimated CIN risk. The CBCIN risk tool estimates CIN risk based on the status of known risk factors (and suggests an associated standard hydration strategy based on left-ventricular end-diastolic pressure), which are automatically prepared from the patient's Electronic Medical Record and presented to the operator for review. This functionality has been evaluated in previous research and was found to be stable and reliable. Based on the data presented by and reviewed in the CBCIN risk tool, the operator may use the information and adjust therapy as clinically indicated (i.e. the risk tool is not the basis for clinical decisions). Following the PCI, serum creatinine will be measured as per treating physician, but those who undergo at least two consecutive daily serum creatinine measurements starting the day after the procedure will be included in the study. These patients will be called 6 months and 12 months post-procedure to determine mortality and re-hospitalization status.

ELIGIBILITY:
Inclusion Criteria:

Inpatients age ≥ 21 years seen at the University of Chicago Medical Center with a clinical indication for cardiac catheterization with high likelihood of PCI, or those undergoing planned PCI will be screened for enrollment into our study. Following PCI, these patients must have at least two consecutive daily creatinine measurements starting the day after the PCI, but clinically-indicated according to the inpatient treating physician.

Exclusion Criteria:

* Patients being discharged the day after the PCI.
* Patients who are screened but do not receive PCI.
* Patients who do not have at least two consecutive daily creatinine measurements starting the day after the PCI.
* Patients undergoing emergency primary percutaneous coronary intervention for ST-segment elevation myocardial infarction.
* Patients in cardiogenic shock.
* Patients with end-stage renal disease or who are on renal replacement therapy.
* Patients requiring planned mechanical circulatory support for the PCI.
* Pregnant women (standard PCI screening)
* Vulnerable populations such as children, college students, prisoners, non-English speakers, and those with diminished decision-making capacity
* Inability or refusal to consent for the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective patient may be considered for the study if they are referred to the University of Chicago Cardiac Catheterization Laboratory as an inpatient for either a planned PCI or a diagnostic angiogram with high likelihood for PCI. For the retrospective control series, subjects will be selected from the electronic medical record starting from the date of the study protocol submission backwards until January 1, 2010 if they meet inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Development of CIN | up to 4 days
  increase in serum creatinine of ≥0.3 mg/dL or ≥50% from the value before the procedure to the highest post-procedure value on days 1-4

CONTACTS AND LOCATIONS:
Overall Officials: John E. A. Blair, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States